CLINICAL TRIAL: NCT06282406
Title: Transcutaneous Auricular Vagus Nerve Stimulation: Motor Learning & Mechanisms
Brief Title: Pupil-Indexed Noninvasive Neuromodulation
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: VA Office of Research and Development (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: N4532-R; I0X1RX004532 (Other Grant/Funding Number: U.S. Department of Veterans Affairs)
Record Dates: First submitted 2024-02-20; First posted 2024-02-28 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: Paresis
Keywords: Learning; Neurological Rehabilitation
MeSH Terms: conditions — Paresis | interventions — Transcutaneous Electric Nerve Stimulation; salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: Subjects will be randomized into one of 5 groups and receive the designated stimulation/sham during a training protocol designed to facilitate motor learning.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (5):
- Paired, Sub-Threshold Stim (Experimental): Sub-threshold stimulation paired with successful task repetitions
  Interventions: Other: Transcutaneous Electrical Stimulation
- Paired, Supra-Threshold Stim (Experimental): Supra-threshold stimulation paired with successful task repetition
  Interventions: Other: Transcutaneous Electrical Stimulation
- Unpaired, Sub-Threshold Stim (Experimental): Sub-threshold stimulation after successful task repetition
  Interventions: Other: Transcutaneous Electrical Stimulation
- Unpaired, Supra-Threshold Stim (Experimental): Supra-threshold stimulation after successful task repetition
  Interventions: Other: Transcutaneous Electrical Stimulation
- Sham (Sham Comparator): No stimulation
  Interventions: Other: Sham

INTERVENTIONS:
Other: Transcutaneous Electrical Stimulation — Electrical pulse trains applied to the skin overlying putative sites of auricular vagal innervation.
  Arms: Paired, Sub-Threshold Stim; Paired, Supra-Threshold Stim; Unpaired, Sub-Threshold Stim; Unpaired, Supra-Threshold Stim
Other: Sham — Electrodes placed on the skin overlying putative sites of auricular vagal innervation but no current administered.
  Arms: Sham

SUMMARY:
Vagus nerve stimulation (VNS) is thought to activate neural pathways that release chemicals which promote plasticity and learning. Previous work has shown that the auricular branch of the vagus nerve innervates landmarks on the external ear. Work from the PI's laboratory has shown that electrical current applied to the external ear modulates physiological indexes of brain states implicated in the therapeutic effects of VNS. The broad objective of this project is to better understand physiological mechanisms modulated by auricular stimulation to support possible therapeutic effects in the form of motor learning.

DETAILED DESCRIPTION:
Existing evidence supports the use of VNS to enhance the effects of traditional therapy on impairments due to neurological injury. It is known that the vagus nerve forms contacts with neuromodulatory nuclei in the brainstem that release of chemicals shown to be critically involved in attentional control and memory formation. It is also known that the auricular branch of the vagus nerve innervates portions of the external ear providing a possible means to engage similar neural pathways noninvasively via transcutaneous auricular vagus nerve stimulation (taVNS). Recent work from the PI's laboratory shows that electrical current applied to landmarks on the external ear elicits transient effects on pupil dilation, an established physiological index of brain states that support learning. Given the ability to engage the biomarker, the investigators aim to further investigate physiological mechanisms modulated by taVNS and possible effects on learning.

ELIGIBILITY:
Inclusion Criteria:

ALL PROSPECTIVE SUBJECTS:

1. 18-75 years of age

   PROSPECTIVE SUBJECTS DIAGNOSED WITH STROKE:
2. Diagnosis of a single stroke resulting in hand impairment
3. Diagnosis of stroke at least six months prior to the time of participation

Exclusion Criteria:

ALL PROSPECTIVE SUBJECTS:

1. History of vestibular disorders or dizziness
2. Difficulty maintaining alertness and/or remaining still
3. Pregnant or expecting to become pregnant
4. Diagnosis of neurological and/or musculoskeletal disorder(s) (other than stroke) that affect movement
5. Ocular disease and/or impairment in more than one eye
6. History of seizure and/or epilepsy
7. Implants, devices, or foreign objects in the brain/body that are incompatible with MRI
8. Body size that is incompatible with MRI scanner dimensions
9. Anyone already enrolled and actively participating in another greater than minimal risk study.

   PROSPECTIVE SUBJECTS DIAGNOSED WITH STROKE:
10. Other impairments secondary to stroke (e.g., attention, cognition, etc.) that would interfere with the ability to understand study goals or follow simple instructions, as judged by the investigators.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 110 (Estimated)
Dates: Start 2024-06-03 (Actual); Primary Completion 2028-04-03 (Estimated); Study Completion 2028-08-05 (Estimated)

PRIMARY OUTCOMES:
Force Control Change | Pre, 1-week Post, 1-month Post
  Subjects will be tested on the same task used for training that involves controlling finger forces.

CONTACTS AND LOCATIONS:
Overall Officials: Michael A. Urbin, PhD, Principal Investigator — VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA
Locations (1):
- VA Pittsburgh Healthcare System University Drive Division, Pittsburgh, PA, Pittsburgh, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dawson J, Liu CY, Francisco GE, Cramer SC, Wolf SL, Dixit A, Alexander J, Ali R, Brown BL, Feng W, DeMark L, Hochberg LR, Kautz SA, Majid A, O'Dell MW, Pierce D, Prudente CN, Redgrave J, Turner DL, Engineer ND, Kimberley TJ. Vagus nerve stimulation paired with rehabilitation for upper limb motor function after ischaemic stroke (VNS-REHAB): a randomised, blinded, pivotal, device trial. Lancet. 2021 Apr 24;397(10284):1545-1553. doi: 10.1016/S0140-6736(21)00475-X. PMID 33894832
- [Background] Follesa P, Biggio F, Gorini G, Caria S, Talani G, Dazzi L, Puligheddu M, Marrosu F, Biggio G. Vagus nerve stimulation increases norepinephrine concentration and the gene expression of BDNF and bFGF in the rat brain. Brain Res. 2007 Nov 7;1179:28-34. doi: 10.1016/j.brainres.2007.08.045. Epub 2007 Aug 25. PMID 17920573
- [Background] Roosevelt RW, Smith DC, Clough RW, Jensen RA, Browning RA. Increased extracellular concentrations of norepinephrine in cortex and hippocampus following vagus nerve stimulation in the rat. Brain Res. 2006 Nov 13;1119(1):124-32. doi: 10.1016/j.brainres.2006.08.048. Epub 2006 Sep 7. PMID 16962076
- [Background] Safi S, Ellrich J, Neuhuber W. Myelinated Axons in the Auricular Branch of the Human Vagus Nerve. Anat Rec (Hoboken). 2016 Sep;299(9):1184-91. doi: 10.1002/ar.23391. Epub 2016 Jul 12. PMID 27342906
- [Background] Butt MF, Albusoda A, Farmer AD, Aziz Q. The anatomical basis for transcutaneous auricular vagus nerve stimulation. J Anat. 2020 Apr;236(4):588-611. doi: 10.1111/joa.13122. Epub 2019 Nov 19. PMID 31742681
- [Background] Urbin MA, Lafe CW, Simpson TW, Wittenberg GF, Chandrasekaran B, Weber DJ. Electrical stimulation of the external ear acutely activates noradrenergic mechanisms in humans. Brain Stimul. 2021 Jul-Aug;14(4):990-1001. doi: 10.1016/j.brs.2021.06.002. Epub 2021 Jun 18. PMID 34154980